CLINICAL TRIAL: NCT06530433
Title: Evaluation of an Enhanced Community First Responder Support System to Improve Bystander Cardiopulmonary Resuscitation Quality for Patients Experiencing Out-of-hospital Cardiac Arrest
Brief Title: Enhanced Community First Responder System Evaluation in Singapore
Acronym: TCPR-Link
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CIRB 2015-2475
Record Dates: First submitted 2024-07-24; First posted 2024-07-31 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: cardiopulmonary resuscitation; Bystander CPR; Community first responder; CPRCard; TCPR Link
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Intervention Model Description: This Health Services research intervention will evaluate effect of live CPR video CPR performance of the volunteer to call-taker in improving CPR Quality and clinical outcomes among the OHCA patients.
Masking Description: Not possible to mask participants and care provider. Outcome is assessed by a device. Analyst will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SoC (Active Comparator): Standard of Care
  Interventions: Device: CPRCard Only
- eCSS (Experimental): enhanced CFR support system (eCSS)
  Interventions: Device: CPRCard + TCPR Link App and Web

INTERVENTIONS:
Device: CPRCard + TCPR Link App and Web — Application that allows responder to perform CPR with two-way audio communication and one-way video streaming to SCDF Dispatcher
  Arms: eCSS
Device: CPRCard Only — Control arm with standard care of procedure that Bystander using CPRCard only
  Arms: SoC

SUMMARY:
The rise in out-of-hospital cardiac arrest (OHCA) cases in Singapore highlights the need for effective bystander cardiopulmonary resuscitation (BCPR). Despite many lay responders performing CPR, survival rates with good neurological outcomes have not significantly improved, prompting research into the quality of CPR as a critical factor. The study by Gallagher EJ et al. showed a significant survival improvement with high-quality CPR.

To address this, the Unit of Pre-hospital and Emergency Research (UPEC) trained thousands of community first responders (CFRs) in simplified CPR techniques using hands-only and DA-CPR methods. A significant innovation is the CPRcard®, developed by Laerdal in Norway, which offers real-time feedback on the quality of chest compressions. However, only 36% of CFRs using the CPRcard® achieved the desired compression standards, indicating room for improvement.

The study proposes enhancing CFR support with information communication technology (ICT), enabling two-way audio and one-way video communication between CFRs and dispatchers. This aims to reduce stress among responders, increase their willingness to engage with OHCA alerts, and improve CPR quality.

The clinical trial in Singapore will compare the current system against the enhanced CFR support system (eCSS), focusing on the real-time relay of CPR performance data, communication ease, and implementation factors. The high-quality CFR and OHCA registries in Singapore provide a robust setting for this research, aiming to enhance CPR delivery and improve OHCA outcomes through technology and real-time support.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above
* SCDF registered CFRs
* Trial dispatchers with an active account of myResponder® app on their mobile phones

Exclusion Criteria:

* The CFRs who are pregnant
* Experiencing any serious physical Conditions
* Mental Health Conditions

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Good Chest Compression Depth (4-6cm) | Throughout chest compression before handing over to EMS (up to 24 hours)
  OHCA events achieving great proportions of adequate compressions (achieving depth within the target range of 4-6 cm)

SECONDARY OUTCOMES:
Survivor discharging rate | Throughout Hospital Admission (up to 1 year)
  Return of spontaneous circulation (ROSC) at scene or at emergency department; survival to discharge; neurologically intact survival

CONTACTS AND LOCATIONS:
Locations (1):
- Duke-NUS Medical School, Singapore, Sigapore, Singapore

REFERENCES:
- [Background] White AE, Ho AF, Shahidah N, Asyikin N, Liew LX, Pek PP, Kua JP, Chia MY, Ng YY, Arulanandam S, Leong SB, Ong ME. An essential review of Singapore's response to out-of-hospital cardiac arrests: improvements over a ten-year period. Singapore Med J. 2021 Aug;62(8):438-443. doi: 10.11622/smedj.2021114. PMID 35001113
- [Background] Ho AFW, Lim MJR, Earnest A, Blewer A, Graves N, Yeo JW, Pek PP, Tiah L, Ong MEH; Singapore PAROS Investigators. Long term survival and disease burden from out-of-hospital cardiac arrest in Singapore: a population-based cohort study. Lancet Reg Health West Pac. 2022 Dec 28;32:100672. doi: 10.1016/j.lanwpc.2022.100672. eCollection 2023 Mar. PMID 36785853
- [Background] Chan PS, McNally B, Tang F, Kellermann A; CARES Surveillance Group. Recent trends in survival from out-of-hospital cardiac arrest in the United States. Circulation. 2014 Nov 18;130(21):1876-82. doi: 10.1161/CIRCULATIONAHA.114.009711. PMID 25399396
- [Background] Gallagher EJ, Lombardi G, Gennis P. Effectiveness of bystander cardiopulmonary resuscitation and survival following out-of-hospital cardiac arrest. JAMA. 1995 Dec 27;274(24):1922-5. PMID 8568985
- [Background] Bobrow BJ, Vadeboncoeur TF, Stolz U, Silver AE, Tobin JM, Crawford SA, Mason TK, Schirmer J, Smith GA, Spaite DW. The influence of scenario-based training and real-time audiovisual feedback on out-of-hospital cardiopulmonary resuscitation quality and survival from out-of-hospital cardiac arrest. Ann Emerg Med. 2013 Jul;62(1):47-56.e1. doi: 10.1016/j.annemergmed.2012.12.020. Epub 2013 Mar 7. PMID 23465553
- [Background] Sasson C, Rogers MA, Dahl J, Kellermann AL. Predictors of survival from out-of-hospital cardiac arrest: a systematic review and meta-analysis. Circ Cardiovasc Qual Outcomes. 2010 Jan;3(1):63-81. doi: 10.1161/CIRCOUTCOMES.109.889576. Epub 2009 Nov 10. PMID 20123673
- [Background] Hollenberg J, Herlitz J, Lindqvist J, Riva G, Bohm K, Rosenqvist M, Svensson L. Improved survival after out-of-hospital cardiac arrest is associated with an increase in proportion of emergency crew--witnessed cases and bystander cardiopulmonary resuscitation. Circulation. 2008 Jul 22;118(4):389-96. doi: 10.1161/CIRCULATIONAHA.107.734137. Epub 2008 Jul 7. PMID 18606920
- [Background] Song J, Guo W, Lu X, Kang X, Song Y, Gong D. The effect of bystander cardiopulmonary resuscitation on the survival of out-of-hospital cardiac arrests: a systematic review and meta-analysis. Scand J Trauma Resusc Emerg Med. 2018 Oct 11;26(1):86. doi: 10.1186/s13049-018-0552-8. PMID 30309373
- [Background] Blewer AL, Ho AFW, Shahidah N, White AE, Pek PP, Ng YY, Mao DR, Tiah L, Chia MY, Leong BS, Cheah SO, Tham LP, Kua JPH, Arulanandam S, Ostbye T, Bosworth HB, Ong MEH. Impact of bystander-focused public health interventions on cardiopulmonary resuscitation and survival: a cohort study. Lancet Public Health. 2020 Aug;5(8):e428-e436. doi: 10.1016/S2468-2667(20)30140-7. PMID 32768435
- [Background] Kim YJ, Ahn S, Sohn CH, Seo DW, Lee YS, Lee JH, Oh BJ, Lim KS, Kim WY. Long-term neurological outcomes in patients after out-of-hospital cardiac arrest. Resuscitation. 2016 Apr;101:1-5. doi: 10.1016/j.resuscitation.2016.01.004. Epub 2016 Jan 28. PMID 26826564
- [Background] White AE, Ng HX, Ng WY, Ng EK, Fook-Chong S, Kua PH, Ong ME. Measuring the effectiveness of a novel CPRcard feedback device during simulated chest compressions by non-healthcare workers. Singapore Med J. 2017 Jul;58(7):438-445. doi: 10.11622/smedj.2017072. PMID 28741006
- [Background] Ong ME, Quah JL, Ho AF, Yap S, Edwin N, Ng YY, Goh ES, Leong BS, Gan HN, Foo DC. National population based survey on the prevalence of first aid, cardiopulmonary resuscitation and automated external defibrillator skills in Singapore. Resuscitation. 2013 Nov;84(11):1633-6. doi: 10.1016/j.resuscitation.2013.05.008. Epub 2013 May 18. PMID 23692983
- [Derived] White AE, Yoon S, Fook-Chong S, Birkenes TS, Ng WM, Naing Win PT, Leong BSH, Jalil NA, Myklebust H, Ong MEH, Siddiqui FJ. Enhanced community first responder support system: protocol of a randomized trial to improve bystander cardiopulmonary resuscitation quality for out-of-hospital cardiac arrest patients. Resusc Plus. 2025 Nov 19;27:101167. doi: 10.1016/j.resplu.2025.101167. eCollection 2026 Jan. PMID 41437946
- See also: Singapore Heart Foundation. Out-of-Hospital Cardiac Arrest Statistics. — https://www.myheart.org.sg/wp-content/uploads/2022/10/Singapore-OHCA-Data-Report-2011-2020.pdf